CLINICAL TRIAL: NCT07141459
Title: Evaluation of the Efficacy of 810 nm Diode Laser Disinfection on Inflammatory Cytokines and Postoperative Pain After Endodontic Retreatment: A Randomized Clinical Trial
Brief Title: Efficacy of 810 nm Diode Laser Disinfection on Inflammatory Cytokines and Postoperative Pain After Endodontic Retreatment
Acronym: cytokines
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Sabah Morad Sobhy, Endodontic department, al azhar university. principal investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P-PD-25-26
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Previous Endodontic Treatment Failure and Radiographically Confirmed Periapical Radiolucency
Keywords: 810 nm diode laser; inflammatory cytokines

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: statician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Diode laser group) (Experimental): Laser activated disinfection will be performed using 810 nm diode laser (Elexxion clarosdental laser, Singen Deutschland, Germany) in a continuous wave mode with a power of 1.5 Watts in 4 cycles of 5 seconds with 20 seconds intervals in between each. Prior to irradiation, all the individuals in the room will wear protective laser safety eye glasses. A 200 μm fiber optic tip (Lite medics, Italy) will be inserted 1 mm from the working length, activated and moved in slow helical motion from the apex to the cervical third with alternating between clockwise and counterclockwise direction at speed of about 2 mm/s(30). 5 ml saline solution will be used for each application and finally before taking post-irradiation sample (S3) using #40 paper points. The teeth will be restored with light cure glass ionomer resin cement temporarily.
  Finally, the root canal system will be obturated using ADSEAL resin-based sealer (Meta Biomed Co, Cheongju, Korea) and gutta-percha.
  Interventions: Device: 810 nm diode laser disinfection
- Group II (Calcium hydroxide group) (Experimental): Calcium hydroxide paste (MetaBiomed, Chungcheongbuk-do, Korea) will be placed inside the root canal and left for 1 week. The access cavity will be temporarily sealed with light cure glass ionomer resin cement. After 1 week, the temporary filling will be removed following local anaesthesia and isolation, the root canal will be irrigated with 20 ml saline and gently filed using H file corresponding to the master apical file size. The last sample (S3) will be collected using #40 paper points. Root canal obturation and final coronal restoration will be completed as in group I
  Interventions: Drug: Calcium Hydroxide Intracanal medication

INTERVENTIONS:
Device: 810 nm diode laser disinfection — 810 nm diode laser (Elexxion clarosdental laser, Singen Deutschland, Germany) in a continuous wave mode with a power of 1.5 Watts in 4 cycles of 5 seconds with 20 seconds intervals in between each. A 200 μm fiber optic tip (Lite medics, Italy) will be inserted 1 mm from the working length, activated and moved in slow helical motion from the apex to the cervical third with alternating between clockwise and counterclockwise direction at speed of about 2 mm/s
  Arms: Group I (Diode laser group)
Drug: Calcium Hydroxide Intracanal medication — Calcium hydroxide paste (MetaBiomed, Chungcheongbuk-do, Korea) will be placed inside the root canal and left for 1 week.
  Arms: Group II (Calcium hydroxide group)

SUMMARY:
The main cause of endodontic disorders is microbial infection. From the infected pulp tissue, microorganisms can penetrate into the deeper layers of root dentine and propagate a periapical tissue through the apical foramen and lateral canals causing apical periodontitis. Apical periodontitis is an inflammatory condition affecting the periapical area of teeth with a global prevalence of 52% among individuals and 5% at tooth level. At the periapical region, microbes and their products encounter the host immune defense. Innate immune cells combat bacteria through phagocytosis and release anti-microbial substances, while adaptive immune cells initiate both cell-mediated and humoral immune responses. This immune activation also stimulates osteoclasts, leading to bone resorption and creating space for the inflammatory cells' infiltration.

During pulpal and periapical inflammation, neutrophils are the predominant immune cells that migrate to the affected area. The main molecules involved in guiding and activating these neutrophils to the site of infection is interleukin-8 (IL-8). This cytokine is locally produced at the site of inflammation and has been linked to pulpal breakdown and apical periodontitis. It promotes the release of tissue-destructive enzymes by neutrophil degranulation. In addition, it affects other leukocyte types such as T cells, B cells, IL-2 activated natural killer cells, and basophils. It has been shown that IL-8 expression is closely related to both infection and inflammation. IL-1β stimulates destruction of periapical tissues which appears to be strongly linked to high microbial load present within the root canal system. It has been identified in teeth exhibiting periapical lesions and root canals containing exudate. Particularly, high levels of IL-1β appear to be related to the presence of clinical signs/ symptoms and destruction of periapical bone Eliminating microorganisms is the primary objective of root canal therapy in order to create an environment as free of bacteria as possible. However, not all root canal treatments are completely successful, and in some cases, the infection persists leading to development of secondary apical periodontitis in previously treated teeth.

Disinfecting the root canal during retreatment is significantly more challenging due to the presence of persistent microorganisms that have settled in the root canal system. These microbes are often resistant to standard irrigations and antimicrobial agents leading to the formation of periradicular lesions. Such bacteria can survive for extended periods around the previously filled root canals. Sodium hypochlorite (NaOCl) is the most widely used irrigant in root canal therapy due to its strong antibacterial effect and its ability to dissolve organic substances. Effective canal cleaning is difficult to achieve without the use of NaOCl at a sufficiently high concentration. However, NaOCl has several drawbacks, including its cytotoxicity which can lead to tissue damage and patient symptoms. Additionally, its strong oxidizing nature negatively affects the mechanical properties of dentin such as microhardness and elastic modulus. NaOCl should be used with caution in endodontic procedures to prevent hypochlorite accidents.

Calcium hydroxide (Ca (OH)2) is the most widely utilized intracanal medication. It has the potential to dissolve tissue, acts as a physical barrier and generates hydroxyl ions, creating an extremely alkaline environment. It has been shown to be quite effective in the treatment of teeth with persistent periapical lesions. To provide optimal endodontic treatment, the root canal system should be thoroughly cleaned of soft-tissue debris, smear layer, and bacteria. However, it is impossible to completely disinfect and clean debris that build up. That is why, adjunctive aids, such as the use of passive ultrasonic and sonic activation of the irrigant and lasers with varying wave lengths, have been introduced during conventional endodontic therapy in cleaning maneuvers.

Laser therapy for root canal disinfection has gained popularity since laser-assisted root canal treatment aims to remove the smear layer, penetrate deep into dentin and eliminate bacteria up to 1000 μm . Laser types have been shown to reduce bacterial load when used as an adjunct to conventional root canal treatment such as Nd:YAG , Er:YAG and diode laser .

DETAILED DESCRIPTION:
Diode laser exhibits a powerful antibacterial effect by altering the bacterial cell wall and damaging the cell membrane. Its photothermal action targets accessible bacteria, while its photodisruptive properties affect those in less accessible areas. This mechanism may not cause immediate bacterial death but instead induces sublethal damage that inhibits bacterial growth. By compromising the integrity of the cell wall and causing the accumulation of denatured proteins, bacterial growth is halted, eventually leading to cell lysis. These effects are achievedwith minimal does of heat.Researches have demonstrated differing degrees of effectiveness in achieving root canal disinfection with the use of diode lasers.

The diode laser is highly well-suited for root canal therapy due to its infrared wavelength and the use of a thin, flexible optic fiber tip (200 µm), which enables deep penetration into the root canal system. This design allows for efficient delivery and distribution of laser energy, improving disinfection and reducing microbial load. Furthermore, the compact size and affordability of diode lasers make them practical for use in general dental clinics and increasing their adoption in routine endodontic procedures. A study demonstrated that 980nm diode laser achieved bactericidal effect ranging from 77 to 97% in root canals infected with E. faecalis using energy outputs of 1.7, 2.3 and 2.8 W. Antimicrobial effect was related to the amount of energy and dentin thickness.

Another study confirmed that the diode laser can serve as an adjunct to conventional root canal therapy in cases with necrotic pulp and periapical radiolucency. Morsy et al evaluated the effectiveness of 980nm diode laser as an adjunctive tool in the retreatment of failed endodontic cases with chronic periapical lesions based on IL-8 expression and postoperative pain, compared to placebo. The findings indicated that intracanal diode laser irradiation is a valuable tool in endodontics, in retreatment cases, contributing to postoperative pain reduction and a decrease in IL-8 expression level.

Postoperative pain is an uncomfortable sensation and a common complication in endodontics, occurring in about 3%-58% of the cases. Pain following root canal obturation can result from various factors including mechanical, chemical or microbial. However; studies have reported that residual microorganisms within the root canal system are the primary contributors, as these microorganisms and byproducts can be extruded to periapical area leading to tissue damage and an increase in the inflammatory mediators' levels.

Although the use of diode laser in root canal disinfection is increasingly common, there is a lack of clinical studies evaluating its biological impact on inflammatory mediators as IL-8 and IL-1β in failed endodontic cases with chronic periapical lesion. Therefore, this study aims to evaluate the impact of 810 nm diode laser on inflammatory cytokines and postoperative pain in endodontic retreatment cases with chronic periapical lesion. The null hypothesis is that there is no difference in the levels of inflammatory cytokines and postoperative pain scores between the diode laser group and calcium hydroxide group following endodontic retreatment

ELIGIBILITY:
Inclusion Criteria:

* Patients have single-rooted teeth with root canal form type I.
* Have previous endodontic therapy with failure.
* Have periapical radiolucency (PAI score of 3 or 4).
* Asymptomatic patients who had no pain or swelling had a negative response to palpation and percussion.
* Patients who provide written informed consent.

Exclusion Criteria:

* Patients who had received antibiotic therapy within the past 3 months. Pregnancy and lactation.
* Systemic disease.
* Physical or mental disability.
* Non restorable teeth.
* Any signs of resorption, immature roots, fracture, sinus tract and dental anomaly

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — cytokine levels varies greatly depending on gender
Enrollment: 52 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-10-20 (Estimated)

PRIMARY OUTCOMES:
IL-8 and IL-1β expression | 1week
  IL-8 and IL-1β levels will be quantified using ELISA kit according to manufacturer instructions

SECONDARY OUTCOMES:
Postoperative pain assessment | • Pre-treatment (baseline). • 6 hours post-treatment. • 12 hours post-treatment. • 1st day post-treatment. • 2nd day post-treatment. • 3rd day post-treatment. • 7th day post-treatment.
  Pain intensity will be assessed using the Visual Analog Scale (VAS) on a 10-point scale (0 = no pain, 10 = worst pain imaginable)

CONTACTS AND LOCATIONS:
Locations (1):
- from the outpatient clinic of Endodontic Department, Faculty of Dental Medicine for Girls, Al-Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morsy DA, Shaker OG, ElKhodary SA. Effect of diode laser (980 nm) on IL-8 expression in failed endodontic cases: Randomised control trial. Aust Endod J. 2025 Apr;51(1):17-25. doi: 10.1111/aej.12914. Epub 2024 Dec 10. PMID 39659152
- [Background] Ozlek E, Kadi G, Shoshaa N, Saed Y, Meydan I. Interleukin-8 (IL-8) levels in gingival crevicular fluid during root canal treatment of molar teeth with symptomatic irreversible pulpitis: impact of varying sodium hypochlorite concentrations. BMC Oral Health. 2024 Mar 27;24(1):392. doi: 10.1186/s12903-024-04128-6. PMID 38539133
- [Background] Tiburcio-Machado CS, Michelon C, Zanatta FB, Gomes MS, Marin JA, Bier CA. The global prevalence of apical periodontitis: a systematic review and meta-analysis. Int Endod J. 2021 May;54(5):712-735. doi: 10.1111/iej.13467. Epub 2021 Jan 22. PMID 33378579